CLINICAL TRIAL: NCT01246206
Title: A Phase II Study of Tacrolimus and Thymoglobulin, as Graft-versus-Host-Disease Prophylaxis in Patients Undergoing Related Donor Hematopoietic Cell Transplantation
Brief Title: Tacrolimus and Thymoglobulin, as GvHD Prophylaxis in Patients Undergoing Related Donor HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSU 2009-095; NCT01414127 (obsolete NCT alias)
Record Dates: First submitted 2010-11-21; First posted 2010-11-23 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Hematological Malignancies
Keywords: ● Non-Hodgkin lymphoma,; ● Hodgkin disease,; ● Acute Myelogenous or Acute Lymphocytic Leukemia; ● Myelodysplastic Syndromes,; ● Chronic Myelogenous Leukemia; ● Multiple Myeloma; ● Chronic Lymphocytic Leukemia; ● Myelofibrosis and other myeloproliferative disorders;
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis | interventions — Tacrolimus; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus and Thymoglobulin (Experimental): Tacrolimus and Thymoglobulin, as Graft-versus-Host-Disease Prophylaxis
  Interventions: Drug: Tacrolimus and Thymoglobulin

INTERVENTIONS:
Drug: Tacrolimus and Thymoglobulin — Intravenous Tacrolimus 0.03 mg/kg/d, beginning day -3, where day 0 is the day of stem cell infusion or "transplant." Intravenous tacrolimus will be discontinued once the participant starts eating, and the drug will then be given orally at a dose of approximately 4 times the intravenous dose. Tacrolimus will be discontinued starting 100 days after transplant unless signs of acute and chronic GVHD develop or if severe toxicity occurs. Thymoglobulin will be given 0.5 mg/kg day-3, Thymoglobulin 1.5 mg/kg day -2, Thymoglobulin 2.5 mg/kg day -1. Thymoglobulin will be given intravenously over 6 hours.
  Other Names: PROGRAF®

SUMMARY:
The primary goal of the study is to determine the incidence and severity of acute Graft versus Host Disease (GVHD) following human leukocyte antigen (HLA) matched related donor Hematopoetic Stem Cell(HSC) transplant in patients with blood related cancers who receive the combination of tacrolimus and Thymoglobulin as GVHD prophylaxis. The investigators also will determine the safety of this combination in the first six months post transplant.

Secondary goals include determining the time to recovery of white blood cells and platelets (engraftment), determining the occurrence of opportunistic infections, defined as infection that occurs in people with weakened immune systems and caused by organisms that do not normally cause disease (fungal infections, pneumocystis carinii pneumonia (PCP), and viral infections), estimating the incidence of chronic GVHD at two years and the overall and disease free survival at two years.

Immune response will be assessed by means of immuno-correlative studies both prior to and at various points after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Suitable related donor as determined by the treating physician
* High resolution molecular HLA typing is mandatory for HLA Class I and II
* Diagnosis of hematological malignancy
* Patients with one of the following hematologic malignancies, and felt to be transplant candidates by their treating physician are eligible to enroll on this protocol:
* Non-Hodgkin lymphoma, any complete remission (CR)/partial remission (PR)
* Hodgkin disease, any CR/PR/stable disease (SD)
* Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) any CR; for non-CR AML or ALL, bone marrow blast < 20% within 4 weeks of transplant and peripheral blood (PB) absolute blast count < 500/μl on the day of initiation of conditioning
* Myelodysplastic syndrome (MDS), treated or untreated
* Chronic myelogenous leukemia (CML) in chronic phase or accelerated phase
* Chronic myelomonocytic leukemia (CMML)
* Multiple myeloma, any CR/PR/SD
* Chronic lymphocytic leukemia (CLL) any CR/PR
* Myelofibrosis and other myeloproliferative disorders; bone marrow blasts less than 20 percent within four weeks of transplant and peripheral blood absolute blast counts less than 500 per microliter on the day of initiation of conditioning
* Age >= 18 and able to cooperate with oral medication intake
* Filgrastim (G-CSF) mobilized Peripheral blood stem cells
* Agrees to participate, and informed consent signed
* Karnofsky performance status (KPS) >= 60, Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Creatinine clearance > 60 mL/min
* Ejection fraction > 50%
* Serum bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST) less than 3 X upper limit of normal
* Forced vital capacity (FVC), forced expiratory volume in one second (FEV1) or diffusion capacity of carbon monoxide (DLCO) > 50% predicted

Exclusion Criteria:

* Bone marrow or Ex vivo engineered or processed graft (cluster of differentiation [CD]34+ enrichment, T-cell depletion, etc)
* Patients with documented uncontrolled central nervous system (CNS) disease
* Active donor or recipient serology positive for human immunodeficiency virus (HIV)
* Known contraindication to administration of Tacrolimus or Thymoglobulin
* Active Hepatitis B or C
* Patients with coronary heart disease (recent myocardial infarctions, angina, cardiac stent, or bypass surgery in the last 6 months) need to be cleared with a stress echocardiogram or nuclear myocardial perfusion stress test, and cardiology consult; all other cardiac history will be at the discretion of the Principal Investigator
* Oxygen usage at the time of enrollment
* Patients with clinical ascites
* Women who are pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus and Thymoglobulin
Started | 21
Completed | 20
Not Completed | 1
Not completed — Patient did not receive study regiments. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 59.5 [38 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute GVHD
Description: Cumulative Incidence of grade II-V acute GVHD with relapse or NRM as competing risks
Time Frame: Assessed first 6 months post transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
percentage of participants | 45.0 [22.3 to 65.4]

2. Primary Outcome: Safety Defined by Serious Adverse Events
Description: Counted the number of participants that experienced any type of grade 3 or higher toxicity.
Time Frame: Assessed first 6 months post transplant
Measure: Number; unit: participants
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
participants | 19

3. Primary Outcome: Severity of Acute GVHD
Description: Cumulative Incidence of grade III-V acute GVHD with relapse or NRM as competing risks
Time Frame: Assessed first 6 months post transplant
Population: Those participants who contracted Acute GVHD
Measure: Number (95% Confidence Interval); unit: % of participants with sever aGVHD
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
% of participants with sever aGVHD | 10.0 [1.6 to 27.8]

4. Secondary Outcome: Determine Incidence of Opportunistic Infections
Time Frame: Followed for up to two years post transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
percentage of participants | 95.0 [75.1 to 99.9]

5. Secondary Outcome: Estimate Incidence of Chronic GVHD at Two Years
Description: Cumulative Incidence of chronic GVHD with relapse or NRM as competing risks
Time Frame: Followed for up to two years post transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
percentage of participants | 75.0 [47.3 to 89.5]

6. Secondary Outcome: Overall Survival at Two Year,
Time Frame: Followed for up to two years post transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
percentage of participants | 75.0 [50.9 to 91.3]

7. Secondary Outcome: Determine Time to Engraftment ("G500")
Description: The number of days until engraftment ("G500")
Time Frame: Followed for up to two years post transplant
Population: All paarticipants
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
days | 11 [7 to 12]

8. Secondary Outcome: Determine Time to Engraftment ("PLT20")
Description: The number of days until engraftment ("PLT20")
Time Frame: Followed for up to two years post transplant
Population: All paarticipants
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus and Thymoglobulin
Number analyzed (Participants) | 20
days | 17 [0 to 25]

ADVERSE EVENTS:
Arm/Group | Tacrolimus and Thymoglobulin
Serious Adverse Events (participants affected / at risk) | 19/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus and Thymoglobulin (N=21)
Alanine Aminotransferase increased (Investigations) | 6 (6)
Aspartate Aminotransferase (AST) (Investigations) | 4 (4)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Asystole (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Bilirubin increase (Investigations) | 4 (4)
Chills (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 5 (5)
Gastric Hemorrhage (Gastrointestinal disorders) | 3 (3)
High cholesterol (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (9)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (11)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypotension (Vascular disorders) | 12 (12)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cytomegalovirus (CMV) infection (Infections and infestations) | 7 (7)
Epstein-Barr virus (EBV) infection (Infections and infestations) | 2 (2)
BK virus infection (Infections and infestations) | 1 (1)
C diff infection (Infections and infestations) | 7 (7)
E coli infection (Infections and infestations) | 3 (3)
E faecalis infection (Infections and infestations) | 1 (1)
Enterococcus raffino infection (Infections and infestations) | 1 (1)
HSV2 Infection (Infections and infestations) | 1 (1)
K oxytoca infection (Infections and infestations) | 1 (1)
Oral candida infection (Infections and infestations) | 1 (1)
Staph coagulase neg (Infections and infestations) | 1 (1)
Staph epi infection (Infections and infestations) | 1 (1)
Staph not aureus (Infections and infestations) | 1 (1)
Strep viridans infection (Infections and infestations) | 2 (2)
TB infection (Infections and infestations) | 1 (1)
UTI infection (Infections and infestations) | 3 (3)
Citrobacter koseri infection (Infections and infestations) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Aspirgillus infection (Infections and infestations) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Gram cocci infection (Infections and infestations) | 2 (2)
Gram neg coccobacil infection (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 8 (8)
Mucositis (Gastrointestinal disorders) | 7 (7)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 12 (12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sinus Tachycardia (Cardiac disorders) | 7 (7)
Syncope (Nervous system disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 2 (2)
Troponin increase (Investigations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Wound infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The small number of patients makes the data hard to interpret.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes